CLINICAL TRIAL: NCT06549283
Title: Nasal Intermittent Positive Pressure Ventilation (NIPPV) During Neonatal Endotracheal Intubation: A Randomized Controlled Trial
Brief Title: Nasal Intermittent Positive Pressure Ventilation During Neonatal Intubation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Muğla Sıtkı Koçman University (Other)
Responsible Party: Principal Investigator, Ozkan Ilhan, Associate Professor, Muğla Sıtkı Koçman University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MSKU-NICU-OI-01
Record Dates: First submitted 2024-08-08; First posted 2024-08-12 (Actual); Last update posted 2024-08-12 (Actual); Status verified 2024-08

CONDITIONS: Respiratory Distress Syndrome; Intubation; Difficult or Failed; Newborn Morbidity; Desaturation of Blood; Ventilator Lung; Newborn
MeSH Terms: conditions — Respiratory Distress Syndrome; Bronchopulmonary Dysplasia

STUDY DESIGN:
Intervention Model Description: The patients were divided into two groups: the NIPPV group and the standard care group.
  In the NIPPV group, NIPPV was implemented during the entire intubation process (pre-intubation to intubation to the end of successful intubation).
  In the standard care group, the intubation attempt proceeded without NIPPV or supplemental oxygen.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- NIPPV group (Active Comparator): Nasal intermittent positive pressure ventilation (NIPPV) was implemented during the entire intubation process (pre-intubation to intubation to the end of successful intubation). Appropriately-sized bi-nasal cannulae were placed prior to laryngoscopy as interface for NIPPV implementation. Non-synchronized NIPPV was implemented. NIPPV was initiated prior to intubation, with the peak inspiratory pressure set to 16-20 cmH2O (selected according to the infant's birth weight and chest wall expansion), positive-end expiratory pressure set to 6 cmH2O, breathing rate set to 40-50 breaths/min, inspiratory time set to 0.40-0.45 s, and flow rate set to 8-12 L/min. After the first successful intubation attempt, NIPPV was discontinued. Prior to laryngoscopy, the fraction of inspired oxygen (FiO2) was adjusted to maintain SpO2 above 90%.
  Interventions: Device: Nasal intermittent positive pressure ventilation (NIPPV) via binasal cannula during neonatal intubation
- Standard-care group (No Intervention): The intubation attempt proceeded without NIPPV or supplemental oxygen.

INTERVENTIONS:
Device: Nasal intermittent positive pressure ventilation (NIPPV) via binasal cannula during neonatal intubation — Researchers applied NIPPV treatment using binasal cannulas through a mechanical ventilator during intubation.
  Arms: NIPPV group

SUMMARY:
The study aims to determine whether the use of nasal intermittent positive pressure ventilation (NIPPV) during neonatal endotracheal intubation increases the rate of successful intubation without physiological instability during all intubation attempts.

The present study was designed as a prospective, multicenter, randomized, controlled study conducted with neonates undergoing endotracheal intubation. The infants were assigned randomly to either the NIPPV group or the standard care group.

DETAILED DESCRIPTION:
The present study was designed as a prospective, multicenter, randomized, controlled trial. The study was conducted at two tertiary Neonatal Intensive Care Units (Mugla Training and Research Hospital, Mugla, Turkey; Akdeniz University School of Medicine, Antalya, Turkey) between May 2023 and May 2024. Written informed consent was obtained from the parents of each neonatal patient prior to enrollment in the study.

Participants:

Infants of a gestational age of 22-41 weeks and undergoing oral endotracheal intubation in the neonatal intensive care unit within the first 28 days of life were eligible for inclusion in the present study. The infants who required urgent intubation, those intubated in the delivery room or the operating room, infants with a heart rate of <120/min prior to randomization, those with airway or lung anomalies, the ones with cyanotic congenital heart disease, and the ones for whom nasal intermittent positive pressure ventilation (NIPPV) treatment was contraindicated (congenital nasal anomaly, congenital diaphragmatic hernia, or abdominal wall defect) were excluded from the study.

Randomization:

Each infant was randomly assigned to either the intervention group or the standard-care group. Sequential numbers were generated in the neonatal intensive care unit's computer with an allocation ratio of 1:1. The numbers were concealed in opaque, sequentially numbered, sealed envelopes. The physician on call opened sequentially numbered sealed opaque envelopes and randomized infants to respective groups before procedure.

Definitions:

An attempt was defined as an airway maneuver, which commenced with the insertion of the laryngoscope blade (conventional) into the mouth of the patient and ended with the removal of the blade. Successful airway management was defined as the placement of an endotracheal tube in the trachea, confirmed based on chest elevation, auscultation, second independent laryngoscopy, carbon dioxide detection, and/or chest radiography. First-attempt success was defined as successful intubation by the first practitioner on the first attempt. Multiple-attempt success was defined as the requirement of over two attempts (≥3) for successful intubation. The requirement for single, two, or multiple attempts for successful intubation was defined as all intubation attempts. Severe oxygen desaturation during intubation was defined as a decrease of ≥20% in oxygen saturation relative to the highest level of oxygen saturation recorded prior to the first attempt. Bradycardia was defined as a heart rate of <100 beats per minute. Physiological instability was defined as severe desaturation (a decrease of >20% in oxygen saturation relative to that immediately prior to pre-laryngoscopy) or bradycardia (a heart rate of <100 beats per minute) during the intubation attempts.

Interventions:

All neonates were monitored using a Philips monitor (IntelliVue MX450) that displayed the real-time peripheral oxygen saturation (SpO2) and heart rate prior to, during, and after the procedure. The patients were divided into two groups: the NIPPV group and the standard care group. In the NIPPV group, NIPPV was implemented during the entire intubation process (pre-intubation to intubation to the end of successful intubation). Appropriately-sized bi-nasal cannulae (Optiflow Junior, Fisher and Paykel, Auckland, New Zealand) were placed prior to laryngoscopy as interface for NIPPV implementation. NIPPV was implemented using Drager Babylog 8000 (Draeger Medicals Inc., Lubeck, Germany) or Leoni Plus (Löwenstein Medical, Bad Ems, Germany) mechanical ventilator. Non-synchronized NIPPV was implemented. NIPPV was initiated prior to intubation, with the peak inspiratory pressure set to 16-20 cmH2O (selected according to the infant's birth weight and chest wall expansion), positive-end expiratory pressure set to 6 cmH2O, breathing rate set to 40-50 breaths/min, inspiratory time set to 0.40-0.45 s, and flow rate set to 8-12 L/min. After the first successful intubation attempt, NIPPV was discontinued. Prior to laryngoscopy, the fraction of inspired oxygen (FiO2) was adjusted to maintain SpO2 above 90%. In the standard care group, the intubation attempt proceeded without NIPPV or supplemental oxygen. In the event of failure in the intubation attempt, SpO2 was increased above 90%, and the heart rate was increased above 120/min by applying positive pressure ventilation using a face mask prior to initiating the next intubation procedure. The size of the intubation tube was determined based on the baby's body weight [12]. Stylet was not used during intubation. Endotracheal intubations were performed either by pediatric research assistants or a neonatologist. A conventional laryngoscope with a straight blade was used for the intubation. Video laryngoscope was not used. Data accuracy was ensured by videotaping the monitor-displayed heart rate and SpO2 during the intubation procedure. After intubation, an independent assessor who was not part of the intubation team reviewed all recorded videos to document the obtained data on a case report form.

Data collection and management:

Data for demographic and clinical characteristics were collected for all patients. A pre-assigned staff member who was not a part of the intubation team noted the vital signs, adverse outcomes, and complications during and after the procedure and also collected blood gas one hour after the intubation for each patient.

Trial outcomes:

The primary outcome was successful intubation without physiological instability during all intubation attempts in the neonate. The secondary outcome was the lowest SpO2 level, lowest heart rate, bradycardia, severe desaturation, duration of severe desaturation, successful intubation on the first attempt without physiological instability, and time to successful intubation.

Sample size:

Hodgson et al. reported that the rate of successful intubation on the first attempt without physiological instability was 31% in newborns who did not receive additional respiratory support during intubation. In the present study, it was hypothesized that the success rate of intubation on the first attempt without physiological instability would increase from 31% to 54% upon the implementation of NIPPV during intubation. The sample size was calculated using the "G*Power 3.1.9.4" program with a type I error of 5% level and a power of 80%. Accordingly, it was concluded that 75 intubation episodes were required for each group, and 150 intubation episodes were required in total.

Statistical analysis:

Statistical analysis was performed using Statistical Package for the Social Sciences (SPSS) software (version 25; Armonk, NY: IBM Corp.). The Kolmogorov-Smirnov and Shapiro-Wilk tests were conducted to determine the normal distribution of data. Student's t-test was conducted to compare the continuous parametric variables. The Mann-Whitney U-test was conducted to compare variables with non-normal distribution. Chi-squared or Fisher's exact test was conducted to analyze the categorical variables. Categorical variables were expressed as numbers (%). Normally distributed variables were expressed as mean ± standard deviation values. Non-parametric continuous variables were expressed as median values (interquartile range). The difference with p < 0.05 was considered statistically significant.

ELIGIBILITY:
Inclusion Criteria:

* Infants of a gestational age of 22-41 weeks and undergoing oral endotracheal intubation in the neonatal intensive care within the first 28 days of life

Exclusion Criteria:

* The infants who required urgent intubation,
* Infants intubated in the delivery room or the operating room,
* Infants with a heart rate of <120/min prior to randomization,
* Infants with airway or lung anomalies,
* Infants with cyanotic congenital heart disease,
* Infants NIPPV treatment was contraindicated (congenital nasal anomaly, congenital diaphragmatic hernia, or abdominal wall defect)

Ages: 1 Day to 28 Days | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 146 (Actual)
Dates: Start 2023-05-01 (Actual); Primary Completion 2024-05-01 (Actual); Study Completion 2024-07-15 (Actual)

PRIMARY OUTCOMES:
Successful intubation without physiological instability during all intubation attempts | One year
  Successful intubation was defined as the placement of an endotracheal tube in the trachea, confirmed based on chest elevation, auscultation, second independent laryngoscopy, carbon dioxide detection, and/or chest radiography.
  Physiological instability was defined as severe desaturation (a decrease of >20% in oxygen saturation relative to that immediately prior to pre-laryngoscopy) or bradycardia (a heart rate of <100 beats per minute) during the intubation attempts.
  All intubation attempts was defined as the requirement for single, two, or multiple attempts for successful intubation.

SECONDARY OUTCOMES:
Lowest SpO2 level | One year
  Lowest peripheral oxygen saturation level during intubation
Lowest heart rate | One year
  Lowest heart rate during intubation
Bradycardia | One year
  Bradycardia was defined as a heart rate of <100 beats per minute
Severe desaturation | One year
  Severe desaturation was defined as a decrease of ≥20% in oxygen saturation relative to the highest level of oxygen saturation recorded prior to the first attempt
Successful intubation on the first attempt without physiological instability | One year
  Successful intubation was defined as the placement of an endotracheal tube in the trachea, confirmed based on chest elevation, auscultation, second independent laryngoscopy, carbon dioxide detection, and/or chest radiography.
  Physiological instability was defined as severe desaturation (a decrease of >20% in oxygen saturation relative to that immediately prior to pre-laryngoscopy) or bradycardia (a heart rate of <100 beats per minute) during the intubation attempts.
Time to successful intubation | One year
  Time until successful intubation is achieved. Successful intubation was defined as the placement of an endotracheal tube in the trachea, confirmed based on chest elevation, auscultation, second independent laryngoscopy, carbon dioxide detection, and/or chest radiography.
Duration of severe desaturation | One year
  Duration of severe desaturation during intubation attempts. Severe desaturation was defined as a decrease of ≥20% in oxygen saturation relative to the highest level of oxygen saturation recorded prior to the first attempt

CONTACTS AND LOCATIONS:
Overall Officials: Ozkan Ilhan, Assoc Prof, Principal Investigator — Muğla Sıtkı Koçman University
Locations (2):
- Turkey (Türkiye) (2):
  - Mugla Training and Research Hospital, Department of Neonatology, Menteşe, Muğla
  - Akdeniz University School of Medicine, Department of Neonatology, Antalya

IPD SHARING:
Plan to Share IPD: No
Our data is available upon request, and we are committed to providing access to interested researchers for the purpose of scientific inquiry.